CLINICAL TRIAL: NCT02369276
Title: Musculoskeletal Ultrasonographic Assessment for the Soft Tissue Injury of Ipsilateral Shoulder of Head and Neck Cancer Patient Following Selective Neck Dissection
Brief Title: Safety Study of Musculoskeletal Ultrasonographic to Assess Disabilities Arm of Head and Neck Cancer Patient
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CMRPG8D1201
Record Dates: First submitted 2015-02-17; First posted 2015-02-23 (Estimated); Last update posted 2018-05-14 (Actual); Status verified 2017-07

CONDITIONS: Head and Neck Cancer
Keywords: neck dissection surgery; shoulder disability; musculoskeletal ultrasonography
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (5):
- post SND within 3 months: 20 Head and Neck Cancer(HNC) complicated with ipsilateral shoulder disability post SND within 3 months, evaluate the soft tissue of shoulder girdle with musculoskeletal ultrasonography and elastography, compare the finding in each group and the range of motion of their shoulder, the severity of wing scapula, visual pain analog scale and the score of The Disability of Arm, Shoulder and Hand
  Interventions: Other: ultrasonography and elastography
- post SND within >3- 6months: 20 Head and Neck Cancer(HNC) complicated with ipsilateral shoulder disability post SND within >3- 6months, evaluate the soft tissue of shoulder girdle with musculoskeletal ultrasonography and elastography, compare the finding in each group and the range of motion of their shoulder, the severity of wing scapula, visual pain analog scale and the score of The Disability of Arm, Shoulder and Hand
  Interventions: Other: ultrasonography and elastography
- post SND within 6 months -1 year: 20 Head and Neck Cancer(HNC) complicated with ipsilateral shoulder disability post SND within 6 months -1 year, evaluate the soft tissue of shoulder girdle with musculoskeletal ultrasonography and elastography, compare the finding in each group and the range of motion of their shoulder, the severity of wing scapula, visual pain analog scale and the score of The Disability of Arm, Shoulder and Hand
  Interventions: Other: ultrasonography and elastography
- post SND within more than 1 year: 20 Head and Neck Cancer(HNC) complicated with ipsilateral shoulder disability post SND within more than 1 year, evaluate the soft tissue of shoulder girdle with musculoskeletal ultrasonography and elastography, compare the finding in each group and the range of motion of their shoulder, the severity of wing scapula, visual pain analog scale and the score of The Disability of Arm, Shoulder and Hand
  Interventions: Other: ultrasonography and elastography
- without shoulder disability: 20 Head and Neck Cancer(HNC) post SND without shoulder complication at the control group, evaluate the soft tissue of shoulder girdle with musculoskeletal ultrasonography and elastography, compare the finding in each group and the range of motion of their shoulder, the severity of wing scapula, visual pain analog scale and the score of The Disability of Arm, Shoulder and Hand
  Interventions: Other: ultrasonography and elastography

INTERVENTIONS:
Other: ultrasonography and elastography — Evaluate the soft tissue of shoulder girdle with musculoskeletal ultrasonography and elastography, compare the finding in each group and the range of motion of their shoulder, the severity of wing scapula, visual pain analog scale and the score of The Disability of Arm, Shoulder and Hand

SUMMARY:
The investigators suppose: 1. SND may cause damage to the soft tissue around shoulder girdle. 2. The soft tissue injury may be related with the order of severity of wing scapula and duration after SND. The aims of this study are: 1. To assess the functional disabilities of shoulder and upper extremity in different time period after SND. 2. To evaluate the soft tissue lesion of shoulder with soft tissue ultrasonography to prove our hypothesis. This study is a two years, prospective, cross-section study. The investigators will enroll 80 HNC post SND within 3months, >3- 6months,> 6months -1 year, more than 1 year as four different groups, 20 patient in each group.

DETAILED DESCRIPTION:
Lymph node metastasis is one the most important prognostic-factors in head and neck cancer(HNC). Radical neck dissection (RND) has been the standard surgical method for HNC with neck lymph nodes metastasis in past decades. This operation includes removal of the sternocleidomastoid muscle (SCM), internal jugular vein (IJV) all cervical lymph nodes on one side and spinal accessory nerve (SAN), leading to significant ipsilateral shoulder syndrome caused by SAN dysfunction and impact quality of life. Despite most clinics prefer to use the nerve-sparing selective neck dissection (SND) for patient with N0 or N1 nodal disease today, shoulder disability and pain were still reported from 31% to 40% after this procedure. However, most previous studies evaluated the shoulder disability only by functional evaluation, range of motion, and questionnaire. The short and long term adverse effect to soft tissue around shoulder girdle after SND has not been reported. The investigators suppose: 1. SND may cause damage to the soft tissue around shoulder girdle. 2. The soft tissue injury may be related with the order of severity of wing scapula and duration after SND. The aims of this study are: 1. To assess the functional disabilities of shoulder and upper extremity in different time period after SND. 2. To evaluate the soft tissue lesion of shoulder with soft tissue ultrasonography to prove our hypothesis. This study is a two years, prospective, cross-section study. The investigators will enroll 80 HNC post SND within 3months, >3- 6months,> 6months -1 year, more than 1 year as four different groups, 20 patient in each group. Evaluate the soft tissue of shoulder girdle with musculoskeletal ultrasonography and elastography, compare the finding in each group and the range of motion of their shoulder, the severity of wing scapula, visual pain analog scale and the score of The Disability of Arm, Shoulder and Hand (DASH) questionnaire. Statistical analysis will perform by SPSS software (SPSS V 20. International Business Machines. USA).

ELIGIBILITY:
Inclusion Criteria:

head and neck cancer by Never-Sparing Selective Neck dissection, SND, the skin condition is stable, there is no wound, infection or inflammation metastasis.

Exclusion Criteria:

(1) in head and neck cancer before surgery and there had been other nerves, bones, muscles, tendons, resulting in lesions of the shoulder pain disorders or a history of activity. (2) severe cognitive function can not meet the examiner. (3) age less than 20 years of age or over 65 years of age.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: head and neck cancer by Never-Sparing Selective Neck dissection, SND, the skin condition is stable, there is no wound, infection or inflammation metastasis. Exclusion criteria: (1) in head and neck cancer before surgery and there had been other nerves, bones, muscles, tendons, resulting in lesions of the shoulder pain disorders or a history of activity. (2) severe cognitive function can not meet the examiner. (3) age less than 20 years of age or over 65 years of age.
Sampling Method: Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2015-04; Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
2-Item findings of musculoskeletal ultrasonography and elastography | baseline

SECONDARY OUTCOMES:
Range of motion | baseline
  Each specific joint has a normal range of motion that is expressed in degrees.Devices to measure range of motion in the joints of the shoulder include the goniometer which use a stationary arm, protractor, fulcrum, and movement arm to measure angle from axis of the joint.
Manual Muscle Test | baseline
  Manual muscle testing is a procedure for the evaluation of the function and strength of individual muscles and muscle groups based on the effective performance of a movement in relation to the forces of gravity and manual resistance.
Pain Scale | baseline
  A pain scale measures a patient's pain intensity or other features. Pain scales are based on self-report, observational (behavioral), or physiological data.
Disabilities of the Arm, Shoulder and Hand questionnaire（DASH） | baseline
  The DASH Outcome Measure is a 30-item, self-report questionnaire designed to measure physical function and symptoms in people with any of several musculoskeletal disorders of the upper limb.

CONTACTS AND LOCATIONS:
Overall Officials: Chau-Peng Leong, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Kaohsiung City, Niaonsung Hsiang, Taiwan

IPD SHARING:
Plan to Share IPD: No
No result now.

REFERENCES:
- [Result] Snow GB, Annyas AA, van Slooten EA, Bartelink H, Hart AA. Prognostic factors of neck node metastasis. Clin Otolaryngol Allied Sci. 1982 Jun;7(3):185-92. doi: 10.1111/j.1365-2273.1982.tb01581.x. PMID 7105450
- [Result] Leemans CR, Tiwari R, Nauta JJ, van der Waal I, Snow GB. Recurrence at the primary site in head and neck cancer and the significance of neck lymph node metastases as a prognostic factor. Cancer. 1994 Jan 1;73(1):187-90. doi: 10.1002/1097-0142(19940101)73:13.0.co;2-j. PMID 8275423
- [Result] Carenfelt C, Eliasson K. Occurrence, duration and prognosis of unexpected accessory nerve paresis in radical neck dissection. Acta Otolaryngol. 1980 Nov-Dec;90(5-6):470-3. doi: 10.3109/00016488009131750. PMID 7211339
- [Result] Hillel AD, Kroll H, Dorman J, Medieros J. Radical neck dissection: a subjective and objective evaluation of postoperative disability. J Otolaryngol. 1989 Feb;18(1):53-61. PMID 2921788
- [Result] Terrell JE, Welsh DE, Bradford CR, Chepeha DB, Esclamado RM, Hogikyan ND, Wolf GT. Pain, quality of life, and spinal accessory nerve status after neck dissection. Laryngoscope. 2000 Apr;110(4):620-6. doi: 10.1097/00005537-200004000-00016. PMID 10764008
- [Result] Gordon SL, Graham WP 3rd, Black JT, Miller SH. Acessory nerve function after surgical procedures in the posterior triangle. Arch Surg. 1977 Mar;112(3):264-8. doi: 10.1001/archsurg.1977.01370030036005. PMID 843216
- [Result] Sobol S, Jensen C, Sawyer W 2nd, Costiloe P, Thong N. Objective comparison of physical dysfunction after neck dissection. Am J Surg. 1985 Oct;150(4):503-9. doi: 10.1016/0002-9610(85)90164-3. PMID 4051117
- [Result] Leipzig B, Suen JY, English JL, Barnes J, Hooper M. Functional evaluation of the spinal accessory nerve after neck dissection. Am J Surg. 1983 Oct;146(4):526-30. doi: 10.1016/0002-9610(83)90246-5. PMID 6625099
- [Result] Short SO, Kaplan JN, Laramore GE, Cummings CW. Shoulder pain and function after neck dissection with or without preservation of the spinal accessory nerve. Am J Surg. 1984 Oct;148(4):478-82. doi: 10.1016/0002-9610(84)90373-8. PMID 6486316
- [Result] El Ghani F, Van Den Brekel MW, De Goede CJ, Kuik J, Leemans CR, Smeele LE. Shoulder function and patient well-being after various types of neck dissections. Clin Otolaryngol Allied Sci. 2002 Oct;27(5):403-8. doi: 10.1046/j.1365-2273.2002.00604.x. PMID 12383306
- [Result] Inoue H, Nibu K, Saito M, Otsuki N, Ishida H, Onitsuka T, Fujii T, Kawabata K, Saikawa M. Quality of life after neck dissection. Arch Otolaryngol Head Neck Surg. 2006 Jun;132(6):662-6. doi: 10.1001/archotol.132.6.662. PMID 16785413
- [Result] Cheng PT, Hao SP, Lin YH, Yeh AR. Objective comparison of shoulder dysfunction after three neck dissection techniques. Ann Otol Rhinol Laryngol. 2000 Aug;109(8 Pt 1):761-6. doi: 10.1177/000348940010900811. PMID 10961810
- [Result] Kuntz AL, Weymuller EA Jr. Impact of neck dissection on quality of life. Laryngoscope. 1999 Aug;109(8):1334-8. doi: 10.1097/00005537-199908000-00030. PMID 10443845
- [Result] Guldiken Y, Orhan KS, Demirel T, Ural HI, Yucel EA, Deger K. Assessment of shoulder impairment after functional neck dissection: long term results. Auris Nasus Larynx. 2005 Dec;32(4):387-91. doi: 10.1016/j.anl.2005.05.007. Epub 2005 Aug 1. PMID 16076539
- [Result] van Wilgen CP, Dijkstra PU, van der Laan BF, Plukker JT, Roodenburg JL. Shoulder and neck morbidity in quality of life after surgery for head and neck cancer. Head Neck. 2004 Oct;26(10):839-44. doi: 10.1002/hed.20052. PMID 15390203
- [Result] van Wouwe M, de Bree R, Kuik DJ, de Goede CJ, Verdonck-de Leeuw IM, Doornaert P, Leemans CR. Shoulder morbidity after non-surgical treatment of the neck. Radiother Oncol. 2009 Feb;90(2):196-201. doi: 10.1016/j.radonc.2008.11.003. Epub 2008 Dec 4. PMID 19054587
- [Result] Tsuji T, Tanuma A, Onitsuka T, Ebihara M, Iida Y, Kimura A, Liu M. Electromyographic findings after different selective neck dissections. Laryngoscope. 2007 Feb;117(2):319-22. doi: 10.1097/01.mlg.0000249781.20989.5c. PMID 17204991
- [Result] Ferlito A, Johnson JT, Rinaldo A, Pratt LW, Fagan JJ, Weir N, Suarez C, Folz BJ, Bien S, Towpik E, Leemans CR, Bradley PJ, Kowalski LP, Herranz J, Gavilan J, Olofsson J. European surgeons were the first to perform neck dissection. Laryngoscope. 2007 May;117(5):797-802. doi: 10.1097/MLG.0b013e3180325b59. PMID 17473671
- [Result] Robbins KT, Medina JE, Wolfe GT, Levine PA, Sessions RB, Pruet CW. Standardizing neck dissection terminology. Official report of the Academy's Committee for Head and Neck Surgery and Oncology. Arch Otolaryngol Head Neck Surg. 1991 Jun;117(6):601-5. doi: 10.1001/archotol.1991.01870180037007. PMID 2036180
- [Result] Brown H, Burns S, Kaiser CW. The spinal accessory nerve plexus, the trapezius muscle, and shoulder stabilization after radical neck cancer surgery. Ann Surg. 1988 Nov;208(5):654-61. doi: 10.1097/00000658-198811000-00019. PMID 3056289
- [Result] Krause HR, Bremerich A, Herrmann M. The innervation of the trapezius muscle in connection with radical neck-dissection. An anatomical study. J Craniomaxillofac Surg. 1991 Feb;19(2):87-9. doi: 10.1016/s1010-5182(05)80613-4. PMID 2037698
- [Result] Patten C, Hillel AD. The 11th nerve syndrome. Accessory nerve palsy or adhesive capsulitis? Arch Otolaryngol Head Neck Surg. 1993 Feb;119(2):215-20. doi: 10.1001/archotol.1993.01880140105016. PMID 8427686
- [Result] Kalra N, Seitz AL, Boardman ND 3rd, Michener LA. Effect of posture on acromiohumeral distance with arm elevation in subjects with and without rotator cuff disease using ultrasonography. J Orthop Sports Phys Ther. 2010 Oct;40(10):633-40. doi: 10.2519/jospt.2010.3155. PMID 20710092
- [Result] Remmler D, Byers R, Scheetz J, Shell B, White G, Zimmerman S, Goepfert H. A prospective study of shoulder disability resulting from radical and modified neck dissections. Head Neck Surg. 1986 Mar-Apr;8(4):280-6. doi: 10.1002/hed.2890080408. PMID 3744856
- [Result] Umeda M, Shigeta T, Takahashi H, Oguni A, Kataoka T, Minamikawa T, Shibuya Y, Komori T. Shoulder mobility after spinal accessory nerve-sparing modified radical neck dissection in oral cancer patients. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2010 Jun;109(6):820-4. doi: 10.1016/j.tripleo.2009.11.027. Epub 2010 Mar 17. PMID 20299249
- [Result] Hudak PL, Amadio PC, Bombardier C. Development of an upper extremity outcome measure: the DASH (disabilities of the arm, shoulder and hand) [corrected]. The Upper Extremity Collaborative Group (UECG). Am J Ind Med. 1996 Jun;29(6):602-8. doi: 10.1002/(SICI)1097-0274(199606)29:63.0.CO;2-L. PMID 8773720
- [Result] Carr SD, Bowyer D, Cox G. Upper limb dysfunction following selective neck dissection: a retrospective questionnaire study. Head Neck. 2009 Jun;31(6):789-92. doi: 10.1002/hed.21018. PMID 19260131
- [Result] Kibler WB, Ludewig PM, McClure PW, Michener LA, Bak K, Sciascia AD. Clinical implications of scapular dyskinesis in shoulder injury: the 2013 consensus statement from the 'Scapular Summit'. Br J Sports Med. 2013 Sep;47(14):877-85. doi: 10.1136/bjsports-2013-092425. Epub 2013 Apr 11. PMID 23580420
- [Result] Grassi W. Clinical evaluation versus ultrasonography: who is the winner? J Rheumatol. 2003 May;30(5):908-9. No abstract available. PMID 12734880
- [Result] Dinnes J, Loveman E, McIntyre L, Waugh N. The effectiveness of diagnostic tests for the assessment of shoulder pain due to soft tissue disorders: a systematic review. Health Technol Assess. 2003;7(29):iii, 1-166. doi: 10.3310/hta7290. PMID 14567906
- [Result] Hawker GA, Mian S, Kendzerska T, French M. Measures of adult pain: Visual Analog Scale for Pain (VAS Pain), Numeric Rating Scale for Pain (NRS Pain), McGill Pain Questionnaire (MPQ), Short-Form McGill Pain Questionnaire (SF-MPQ), Chronic Pain Grade Scale (CPGS), Short Form-36 Bodily Pain Scale (SF-36 BPS), and Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S240-52. doi: 10.1002/acr.20543. No abstract available. PMID 22588748
- [Result] Martin RM, Fish DE. Scapular winging: anatomical review, diagnosis, and treatments. Curr Rev Musculoskelet Med. 2008 Mar;1(1):1-11. doi: 10.1007/s12178-007-9000-5. PMID 19468892
- [Result] Ophir J, Cespedes I, Ponnekanti H, Yazdi Y, Li X. Elastography: a quantitative method for imaging the elasticity of biological tissues. Ultrason Imaging. 1991 Apr;13(2):111-34. doi: 10.1177/016173469101300201. PMID 1858217
- [Result] Righetti R, Garra BS, Mobbs LM, Kraemer-Chant CM, Ophir J, Krouskop TA. The feasibility of using poroelastographic techniques for distinguishing between normal and lymphedematous tissues in vivo. Phys Med Biol. 2007 Nov 7;52(21):6525-41. doi: 10.1088/0031-9155/52/21/013. Epub 2007 Oct 16. PMID 17951860
- [Result] Varghese T, Ophir J. Performance optimization in elastography: multicompression with temporal stretching. Ultrason Imaging. 1996 Jul;18(3):193-214. doi: 10.1177/016173469601800303. PMID 9123673
- [Result] Drakonaki EE, Allen GM, Wilson DJ. Ultrasound elastography for musculoskeletal applications. Br J Radiol. 2012 Nov;85(1019):1435-45. doi: 10.1259/bjr/93042867. PMID 23091287
- [Result] Grainger AJ. Highlights of the European Society of Musculoskeletal Radiology (ESSR) annual meeting 2010. Skeletal Radiol. 2011 Jan;40(1):137-9. doi: 10.1007/s00256-010-1030-1. No abstract available. PMID 21104049